CLINICAL TRIAL: NCT04116229
Title: Neuroinflammation in Obesity
Brief Title: Cognition and Magnetic Resonance Imaging of Brain Inflammation in Obesity
Acronym: NIFOB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Sarah Eisenstein, Assistant Professor, Washington University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: 201805053; P30DK020579 (NIH)
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Results first posted 2022-10-19 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Obesity
Keywords: Obesity; Inflammation; Cognitive impairment; Neuroimaging; Magnetic resonance imaging
MeSH Terms: conditions — Obesity; Inflammation; Cognitive Dysfunction | interventions — Glucose Tolerance Test; Neuropsychological Tests; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: This study employed a single group model in which participants with obesity and participants with normal-weight underwent magnetic resonance imaging, blood draws and cognitive assessment.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Neuroimaging data was processed using automated methods blind to group membership. Blood samples were analyzed by laboratory personnel blind to group membership.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal-weight (Active Comparator): Participants who have a body mass index within the normal-weight category.
  Interventions: Procedure: Oral glucose tolerance test; Behavioral: Cognitive testing; Procedure: Magnetic resonance imaging
- Obese (Active Comparator): Participants who have a body mass index within the obese category.
  Interventions: Procedure: Oral glucose tolerance test; Behavioral: Cognitive testing; Procedure: Magnetic resonance imaging

INTERVENTIONS:
Procedure: Oral glucose tolerance test — After 8 hours fasting overnight, an intravenous catheter is placed in the arm or hand for blood draws. Participants drink 75 grams of an oral glucose drink after baseline blood samples are drawn. More blood draws occur at 10, 20, 30, 60 and 120 min post-glucose drink.
Behavioral: Cognitive testing — For approximately 40 minutes, participants are assessed for cognitive function using computer-based tests available from the NIH Toolbox Cognitive Battery (Weintraub et al., 2013), including attention and executive functioning, episodic memory, working memory, language, processing speed, and immediate recall.
Procedure: Magnetic resonance imaging — Magnetic resonance imaging (MRI) scans will be performed in a 3 Tesla MRI scanner over 1.5 hours. Participants will be asked to lay down flat on their backs and to try to stay still throughout the MRI scan. The participant will wear MRI-safe headphones to block out noise due to the MRI scans. Participant comfort will be verbally checked on throughout the scan and the participant will be provided with a 'squeeze ball' to signal the MRI technician that they want to get out of the scanner immediately.

SUMMARY:
The rate of obesity in the United States is high and is a risk factor for concurrent cognitive impairment and, in late life, dementias such as Alzheimer's disease. In order to prevent or reduce cognitive impairment, the mechanism underlying the link between obesity and cognitive impairment must be understood. The current study aims to provide preliminary data on whether brain inflammation occurs in obesity and relates to cognitive deficits using magnetic resonance neuroimaging and cognitive testing. It is hypothesized that obese individuals will have greater brain inflammation and lower cognitive function compared to normal-weight individuals. Further, it is predicted that brain inflammation will relate to cognitive function and plasma indicators of inflammation in obese individuals.

DETAILED DESCRIPTION:
Initially, normal-weight or obese potential participants are screened by a phone interview that assesses medical history. Obtainment of informed consent and further screening occurs on the day of the study visit. Participants then undergo a 2 hour oral glucose tolerance test (OGTT) including blood draws for metabolic and inflammatory marker levels in plasma. Lunch is then provided. Participants are then administered 30 minute computer-based cognitive testing from the NIH Toolbox Cognition Battery. After cognitive testing, participants undergo 1.5 hour magnetic resonance imaging (MRI) that includes structural, diffusion tensor, and functional MR imaging.

ELIGIBILITY:
Inclusion Criteria:

* Non-obese (body mass index = 18 - 25 kg/m^2) or Obese (body mass index ≥ 30 kg/m^2
* Any race or ethnicity
* Native English speaker

Exclusion Criteria:

* Past or current diabetes
* Current psychotropic medication use
* Past or current neurological illness
* Past or current substance or alcohol misuse
* Past or current mental illness
* Current binge eating disorder
* Magnetic resonance imaging contraindications
* Pregnancy
* Currently lactating
* Tobacco use within past month
* Over 350 lb

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Hershey, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data is available immediately as of August 15, 2022 for 5 years.
Access Criteria: Upon reasonable request

REFERENCES:
- [Background] Weintraub S, Dikmen SS, Heaton RK, Tulsky DS, Zelazo PD, Bauer PJ, Carlozzi NE, Slotkin J, Blitz D, Wallner-Allen K, Fox NA, Beaumont JL, Mungas D, Nowinski CJ, Richler J, Deocampo JA, Anderson JE, Manly JJ, Borosh B, Havlik R, Conway K, Edwards E, Freund L, King JW, Moy C, Witt E, Gershon RC. Cognition assessment using the NIH Toolbox. Neurology. 2013 Mar 12;80(11 Suppl 3):S54-64. doi: 10.1212/WNL.0b013e3182872ded. PMID 23479546
- [Background] Cross AH, Song SK. "A new imaging modality to non-invasively assess multiple sclerosis pathology". J Neuroimmunol. 2017 Mar 15;304:81-85. doi: 10.1016/j.jneuroim.2016.10.002. Epub 2016 Oct 8. PMID 27773433
- [Background] Breda E, Cavaghan MK, Toffolo G, Polonsky KS, Cobelli C. Oral glucose tolerance test minimal model indexes of beta-cell function and insulin sensitivity. Diabetes. 2001 Jan;50(1):150-8. doi: 10.2337/diabetes.50.1.150. PMID 11147781
- See also: NIH Toolbox Cognitive Battery description — http://www.healthmeasures.net/explore-measurement-systems/nih-toolbox/intro-to-nih-toolbox/cognition

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normal-weight | Obese
Started | 10 | 10
Completed | 8 | 6
Not Completed | 2 | 4
Not completed — Met exclusion criteria during screeneing on day of study visit. | 2 | 3
Not completed — Scheduling not possible. | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal-weight | Obese | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (6.6) | 36.5 (6.8) | 35.6 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black, non-Hispanic | 1 | 2 | 3
  White, non-Hispanic | 6 | 4 | 10
  Asian, non-Hispanic | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 6 | 14
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 22.4 (1.5) | 37.3 (4.5) | 28.7 (8.2)
HbA1c [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 5.1 (0.1) | 5.1 (0.4) | 5.1 (0.2)
Fasting glucose [Mean (Standard Deviation); unit: mg/dL] | 87.0 (4.6) | 87.2 (8.0) | 87.0 (6.0)
Fasting plasma insulin [Mean (Standard Deviation); unit: uU/mL] | 5.28 (3.73) | 15.62 (10.82) | 9.71 (9.0)
Homeostatic measure of insulin resistance (HOMA-IR) [Mean (Standard Deviation); unit: unitless] — Homeostatic model for insulin resistance, where greater HOMA-IR indicates greater insulin resistance.
  unitless | 1.21 (0.79) | 3.47 (2.56) | 2.18 (2.05)
Fasting plasma free fatty acid (FFA) [Mean (Standard Deviation); unit: mEq/L] | 0.61 (0.27) | 0.81 (0.29) | 0.7 (0.29)
Fasting plasma C-reactive protein (CRP) [Mean (Standard Deviation); unit: mg/L] — Pro-inflammatory marker
  mg/L | 1.02 (0.8) | 4.84 (3.1) | 2.66 (2.8)
Fasting plasma monocyte chemoattractant protein-1 (MCP-1) [Mean (Standard Deviation); unit: pg/mL] — Pro-inflammatory marker
  pg/mL | 140.9 (37.0) | 160.3 (40.1) | 149.2 (38.2)
Fasting plasma tumor necrosis factor-alpha (TNF-alpha) [Mean (Standard Deviation); unit: pg/mL] — Pro-inflammatory marker
  pg/mL | 0.69 (0.16) | 0.84 (0.16) | 0.75 (0.17)
Fasting plasma adiponectin [Mean (Standard Deviation); unit: ug/mL] — Anti-inflammatory marker
  ug/mL | 11.3 (5.6) | 10.8 (4.9) | 11.1 (5.1)
Fasting plasma interleukin-10 (IL-10) [Mean (Standard Deviation); unit: pg/mL] — Anti-inflammatory marker
  pg/mL | 1.85 (1.38) | 1.97 (0.75) | 1.9 (1.12)
Fasting plasma leptin [Mean (Standard Deviation); unit: ug/L] — "Satiety" hormone
  ug/L | 19.9 (13.4) | 110 (49.7) | 58.5 (56.4)
Fasting plasma ghrelin [Mean (Standard Deviation); unit: pg/mL] — "Hunger" hormone
  pg/mL | 1498.5 (568.6) | 914.8 (261.7) | 1248.4 (538.8)

OUTCOME MEASURES:

1. Primary Outcome: Brain Inflammation Metrics in Obese and Normal-weight Individuals as Measured by Magnetic Resonance Image-based Diffusion Basis Spectrum Imaging (DBSI)
Description: Diffusion Basis Spectrum Imaging (Cross and Song, 2017) is a computational method that will be applied to diffusion tensor images of the brain to estimate putative inflammation-related markers including cellularity and edema in obese and normal-weight individuals. DBSI metrics are quantitative but unitless. Cellularity and edema fractions of the total diffusion signal (including axial, radial, restricted (cellularity) and hindered (edema)) will be estimated in brain white matter tracts.
Time Frame: 1.5 hours at the end of one (up to) 8 hour study day that includes all outcome measures
Population: Data from 8 individuals with normal-weight and 6 individuals with obesity were included in baseline analyses. Five individuals were enrolled in the study but their data was not collected due to meeting exclusion criteria. One individual was enrolled but could not be scheduled for the study and therefore did not contribute data.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Normal-weight | Obese
Number analyzed (Participants) | 8 | 6
unitless
  DBSI restricted fraction (cellularity) | .0468 (.0024) | .0492 (.0034)
  DBSI hindered fraction (vasogenic edema) | .176 (.013) | .186 (.014)
Statistical Analysis 1: Comparison: Normal-weight vs Obese; This is a pilot study with a small sample. Power to detect significant results is therefore low in the current study; Test type: Equivalence — Alternative hypothesis: people with normal-weight BMI have lower DBSI restricted fraction, or putative cellularity, than people with obesity. Null hypothesis: DBSI restricted fraction, or putative cellularity, is not different between normal-weight and obese groups; p = 0.28, Independent-Samples Median Test — a priori threshold: p < 0.05; Median Difference (Final Values) = 0.05
Statistical Analysis 2: Comparison: Normal-weight vs Obese; This is a pilot study with a small sample. Power to detect significant results is therefore low in the current study; Test type: Equivalence — Alternative hypothesis: people with normal-weight BMI have lower DBSI hindered fraction, or putative vasogenic edema, than people with obesity. Null hypothesis: DBSI hindered fraction, or putative vasogenic edema, is not different between normal-weight and obese groups; p = 0.03, Independent-Samples Median Test — a priori threshold: p < 0.05; Median Difference (Final Values) = 0.18

2. Primary Outcome: Cognitive Function in Obese and Normal-weight Individuals as Measured by the National Institutes of Health (NIH) Toolbox Cognitive Battery and DBSI Putative Neuroinflammation Metrics
Description: Cognitive performance including fluid and crystallized cognition composite T-scores from computer-based NIH Cognitive Toolbox assessments (Weintraub et al., 2013) will be assessed in obese and normal-weight individuals. These T-scores will include scores from tasks that assess attention and executive functioning, episodic memory, working memory, language, processing speed, and immediate recall (see NIH Toolbox Cognitive Battery website). T-scores are corrected for socioeconomic status and their distribution has a mean of 50 and a standard deviation of 10. Higher T-scores indicate better cognitive function. T-scores will be correlated with DBSI-assessed neuroinflammation metrics including restricted fraction (DBSI RF, putative cellularity) and hindered fraction (DBSI HF, putative vasogenic edema) in brain white matter tracts.
Time Frame: 40 minutes during one (up to) 8 hour study day that includes all outcome measures; after OGTT and prior to MRI
Population: Two individuals in the normal-weight group were not native English speakers and their cognitive data is not included. A complete set of fluid cognition measures was not collected from one normal-weight participant and their fluid cognition data is not included.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Normal-weight | Obese
Number analyzed (Participants) | 6 | 6
T-score
  Crystallized Cognition | 60.3 (6.9) | 53.3 (9.0)
  Fluid Cognition: number analyzed (Participants) | 5 | 6
  Fluid Cognition | 54.4 (6.7) | 59.3 (7.4)
Statistical Analysis 1: Comparison: Normal-weight vs Obese; This is a pilot study with a small sample. Power to detect significant results is therefore low in the current study. Analyses performed across normal-weight and obese groups; Test type: Other — Alternative hypothesis: Worse crystallized cognitive function will relate to greater putative vasogenic edema (DBSI HF) in white matter tracts. Null hypothesis: Crystallized cogntive function is not related to DBSI HF; p = 0.01, Regression, Linear — a priori threshold: p < 0.05; Slope = -0.69
Statistical Analysis 2: Comparison: Normal-weight vs Obese; [analysis description as in outcome 2, analysis 1]; Test type: Other — Alternative hypothesis: Worse fluid cognitive function will relate to greater putative vasogenic edema (DBSI HF) in white matter tracts. Null hypothesis: Fluid cogntive function is not related to DBSI HF; p = 0.10, Regression, Linear — a priori threshold: p < 0.05; Slope = 0.52
Statistical Analysis 3: Comparison: Normal-weight vs Obese; [analysis description as in outcome 2, analysis 1]; Test type: Other — Alternative hypothesis: Worse crystallized cognitive function will relate to greater putative cellularity (DBSI RF) in white matter tracts. Null hypothesis: Crystallized cognitive function is not related to DBSI RF; p = 0.01, Regression, Linear — a priori threshold: p < 0.05; Slope = -0.45
Statistical Analysis 4: Comparison: Normal-weight vs Obese; [analysis description as in outcome 2, analysis 1]; Test type: Other — Alternative hypothesis: Worse fluid cognitive function will relate to greater putative cellularity (DBSI RF) in white matter tracts. Null hypothesis: Fluid cognitive function is not related to DBSI RF; p = 0.10, Regression, Linear — a priori threshold: p < 0.05; Slope = 0.22

3. Post Hoc Outcome: Metabolic Markers in Plasma and Relationships With DBSI Neuroinflammation Metrics in White Matter Tracts in Obese and Normal-weight Individuals.
Description: Fasting plasma insulin, a measure of insulin resistance in which higher levels may reflect greater effort to maintain glucose homeostasis, was measured by radioimmunoassay. Normal fasting plasma insulin levels are < 25 uU/mL.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: uU/mL
Arm/Group | Normal-weight | Obese
Number analyzed (Participants) | 8 | 6
uU/mL | 5.28 (3.73) | 15.62 (10.82)
Statistical Analysis 1: Comparison: Normal-weight vs Obese; [analysis description as in outcome 2, analysis 1]; Test type: Other — Alternative hypothesis: higher levels of insulin, a pro-inflammatory marker, will relate to higher levels of putative neuroinflammation in white matter tracts as measured by DBSI restricted fraction after controlling for BMI. Null hypothesis: Insulin levels will not be related to DBSI RF in white matter tracts after controlling for BMI; p > 0.46, Regression, Linear — a priori threshold: p < 0.05; Slope = -0.18
Statistical Analysis 2: Comparison: Normal-weight vs Obese; [analysis description as in outcome 2, analysis 1]; Test type: Other — Alternative hypothesis: higher levels of insulin, a pro-inflammatory marker, will relate to higher levels of putative neuroinflammation in white matter tracts as measured by DBSI hindered fraction after controlling for BMI. Null hypothesis: Insulin levels will not be related to DBSI HF in white matter tracts after controlling for BMI; p > 0.5, Regression, Linear — a priori threshold: p < 0.05; Slope = -0.22

4. Post Hoc Outcome: Metabolic Markers in Plasma and Relationships With DBSI Neuroinflammation Metrics in White Matter Tracts in Obese and Normal-weight Individuals.
Description: Fasting plasma leptin, a hormone related to adipose tissue mass such that higher levels reflect greater adipose tissue mass, was measured by radioimmunoassay.
  For body mass index (BMI) in normal-weight (18.5-24.9 kg/m^2), leptin reference range = 1.8-24.2 ug/L in females and 0.2-7.7 in males. For BMI in individuals with obesity, leptin reference range = 10.6-141 in females and 3.2-135 in males.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Normal-weight | Obese
Number analyzed (Participants) | 8 | 6
ug/L | 19.9 (13.4) | 110 (49.7)
Statistical Analysis 1: Comparison: Normal-weight vs Obese; [analysis description as in outcome 2, analysis 1]; Test type: Other — Alternative hypothesis: higher levels of leptin, a pro-inflammatory marker and "satiety" hormone, will relate to higher levels of putative neuroinflammation in white matter tracts as measured by DBSI restricted fraction after controlling for BMI. Null hypothesis: Leptin levels will not be related to DBSI RF in white matter tracts after controlling for BMI; p = 0.62, Regression, Linear — a priori threshold: p < 0.05; Slope = 0.15
Statistical Analysis 2: Comparison: Normal-weight vs Obese; [analysis description as in outcome 2, analysis 1]; Test type: Other — Alternative hypothesis: higher levels of leptin, a pro-inflammatory marker and "satiety" hormone, will relate to higher levels of putative neuroinflammation in white matter tracts as measured by DBSI hindered fraction after controlling for BMI. Null hypothesis: Leptin levels will not be related to DBSI HF in white matter tracts after controlling for BMI; p = 0.82, Regression, Linear; Slope = -0.07

5. Post Hoc Outcome: Metabolic Markers in Plasma and Relationships With DBSI Neuroinflammation Metrics in White Matter Tracts in Obese and Normal-weight Individuals.
Description: Fasting plasma ghrelin, a hormone related to hunger in which higher levels may signal the stomach is empty and it is time to eat, was measured by radioimmunoassay.
  Plasma ghrelin levels tend to be lower in people with obesity. There is no established normal range for fasting plasma ghrelin levels as assessed by radioimmunoassay.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Normal-weight | Obese
Number analyzed (Participants) | 8 | 6
pg/mL | 1498.5 (568.6) | 914.8 (261.7)
Statistical Analysis 1: Comparison: Normal-weight vs Obese; [analysis description as in outcome 2, analysis 1]; Test type: Other — Alternative hypothesis: higher levels of ghrelin, an anti-inflammatory marker and "hunger" hormone, will relate to lower levels of putative neuroinflammation in white matter tracts as measured by DBSI restricted fraction after controlling for BMI. Null hypothesis: Ghrelin levels will not be related to DBSI RF in white matter tracts after controlling for BMI; p = 0.53, Regression, Linear — a priori threshold: p < 0.05; Slope = 0.19
Statistical Analysis 2: Comparison: Normal-weight vs Obese; [analysis description as in outcome 2, analysis 1]; Test type: Other — Alternative hypothesis: higher levels of ghrelin, an anti-inflammatory marker and "hunger" hormone, will relate to lower levels of putative neuroinflammation in white matter tracts as measured by DBSI hindered fraction after controlling for BMI. Null hypothesis: Ghrelin levels will not be related to DBSI HF in white matter tracts after controlling for BMI; p = 0.71, Regression, Linear — a priori threshold: p < 0.05; Slope = -0.12

6. Post Hoc Outcome: Metabolic Markers in Plasma and Relationships With DBSI Neuroinflammation Metrics in White Matter Tracts in Obese and Normal-weight Individuals.
Description: Homeostatic measure of insulin resistance (HOMA-IR) where higher scores indicate greater insulin resistance, or diminished maintenance of glucose homeostasis by insulin. HOMA-IR was calculated according to the formula: fasting insulin (uU/L) * fasting glucose (nmol/L)/22.5
  A HOMA-IR score >2.5 indicates insulin resistance.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: HOMA-IR score
Arm/Group | Normal-weight | Obese
Number analyzed (Participants) | 8 | 6
HOMA-IR score | 1.21 (0.79) | 3.47 (2.56)
Statistical Analysis 1: Comparison: Normal-weight vs Obese; [analysis description as in outcome 2, analysis 1]; Test type: Other — Alternative hypothesis: greater HOMA-IR, where higher HOMA-IR indicates greater insulin resistance, will relate to higher levels of putative neuroinflammation in white matter tracts as measured by DBSI restricted fraction after controlling for BMI. Null hypothesis: HOMA-IR levels will not be related to DBSI RF in white matter tracts after controlling for BMI; p = 0.53, Regression, Linear — a priori threshold: p < 0.05; Slope = -0.19
Statistical Analysis 2: Comparison: Normal-weight vs Obese; [analysis description as in outcome 2, analysis 1]; Test type: Other — Alternative hypothesis: greater HOMA-IR, where higher HOMA-IR indicates greater insulin resistance, will relate to higher levels of putative neuroinflammation in white matter tracts as measured by DBSI hindered fraction after controlling for BMI. Null hypothesis: HOMA-IR levels will not be related to DBSI HF in white matter tracts after controlling for BMI; p = 0.5, Regression, Linear; Slope = -0.21

7. Post Hoc Outcome: Peripheral Inflammation as Measured by Plasma Assays and Relationships With DBSI Putative Neuroinflammation Metrics in White Matter Tracts in Obese and Normal-weight Individuals
Description: Fasting plasma interleukin (IL)-10, an anti-inflammatory cytokine important for immune response. IL-10 was measured using high-sensitive enzyme-linked immuno-absorbent assay (ELISA). Normal reference ranges for IL-10 have not been established and better or worse levels depend on disease state.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Normal-weight | Obese
Number analyzed (Participants) | 8 | 6
pg/mL | 1.85 (1.38) | 1.97 (0.75)
Statistical Analysis 1: Comparison: Normal-weight vs Obese; [analysis description as in outcome 2, analysis 1]; Test type: Other — Alternative hypothesis: higher levels of IL-10, an anti-inflammatory marker, will relate to lower levels of putative neuroinflammation in white matter tracts as measured by DBSI restricted fraction after controlling for BMI. Null hypothesis: IL-10 levels will not be related to DBSI RF in white matter tracts after controlling for BMI; p = 0.09, Regression, Linear — a priori threshold: p < 0.05; Slope = 0.5
Statistical Analysis 2: Comparison: Normal-weight vs Obese; [analysis description as in outcome 2, analysis 1]; Test type: Other — Alternative hypothesis: higher levels of IL-10, an anti-inflammatory marker, will relate to lower levels of putative neuroinflammation in white matter tracts as measured by DBSI hindered fraction after controlling for BMI. Null hypothesis: IL-10 levels will not be related to DBSI HF in white matter tracts after controlling for BMI; p = 0.45, Regression, Linear — a priori threshold: p < 0.05; Slope = -0.2

8. Post Hoc Outcome: Peripheral Inflammation as Measured by Plasma Assays and Relationships With DBSI Putative Neuroinflammation Metrics in White Matter Tracts in Obese and Normal-weight Individuals
Description: Fasting plasma adiponectin, an anti-inflammatory cytokine important for immune response. Adiponectin was measured using radioimmunoassay. Normal reference ranges for adiponectin is 2.5-21.1 ug/mL. Lower levels of adiponectin tend to be associated with worse metabolic health and higher body mass index.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Normal-weight | Obese
Number analyzed (Participants) | 8 | 6
ug/mL | 11.3 (5.6) | 10.8 (4.9)
Statistical Analysis 1: Comparison: Normal-weight vs Obese; [analysis description as in outcome 2, analysis 1]; Test type: Other — Alternative hypothesis: higher levels of adiponectin, an anti-inflammatory marker, will relate to lower levels of putative neuroinflammation in white matter tracts as measured by DBSI restricted fraction after controlling for BMI. Null hypothesis: Adiponectin levels will not be related to DBSI RF in white matter tracts after controlling for BMI; p = 0.19, Regression, Linear — a priori threshold: p < 0.05; Slope = 0.38
Statistical Analysis 2: Comparison: Normal-weight vs Obese; [analysis description as in outcome 2, analysis 1]; Test type: Other — Alternative hypothesis: higher levels of adiponectin, an anti-inflammatory marker, will relate to lower levels of putative neuroinflammation in white matter tracts as measured by DBSI hindered fraction after controlling for BMI. Null hypothesis: Adiponectin levels will not be related to DBSI HF in white matter tracts after controlling for BMI; p = 0.52, Regression, Linear — a priori threshold: p < 0.05; Slope = -0.2

9. Post Hoc Outcome: Peripheral Inflammation as Measured by Plasma Assays and Relationships With DBSI Putative Neuroinflammation Metrics in White Matter Tracts in Obese and Normal-weight Individuals
Description: Fasting plasma tumor necrosis factor (TNF)-alpha, a pro-inflammatory cytokine important for systemic inflammation. TNF-alpha was measured using high-sensitive enzyme-linked immuno-absorbent assay (ELISA). Normal TNF-alpha levels range from non-detectable to 8.1 pg/mL and tend to be higher in people with obesity compared to normal-weight.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Normal-weight | Obese
Number analyzed (Participants) | 8 | 6
pg/mL | 0.69 (0.16) | 0.84 (0.16)
Statistical Analysis 1: Comparison: Normal-weight vs Obese; [analysis description as in outcome 2, analysis 1]; Test type: Other — Alternative hypothesis: higher levels of TNF-alpha, a pro-inflammatory marker, will relate to higher levels of putative neuroinflammation in white matter tracts as measured by DBSI restricted fraction after controlling for BMI. Null hypothesis: TNF-alpha levels will not be related to DBSI RF in white matter tracts after controlling for BMI; p = 0.90, Regression, Linear — a priori threshold: p < 0.05; Slope = -0.05
Statistical Analysis 2: Comparison: Normal-weight vs Obese; [analysis description as in outcome 2, analysis 1]; Test type: Other — Alternative hypothesis: higher levels of TNF-alpha, a pro-inflammatory marker, will relate to higher levels of putative neuroinflammation in white matter tracts as measured by DBSI hindered fraction after controlling for BMI. Null hypothesis: TNF-alpha levels will not be related to DBSI HF in white matter tracts after controlling for BMI; p = 0.87, Regression, Linear — a priori threshold: p < 0.05; Slope = 0.04

10. Post Hoc Outcome: Peripheral Inflammation as Measured by Plasma Assays and Relationships With DBSI Putative Neuroinflammation Metrics in White Matter Tracts in Obese and Normal-weight Individuals
Description: Fasting plasma monocyte chemoreactant protein (MCP)-1, a pro-inflammatory chemokine important for immune response and inflammation. MCP-1 was measured using enzyme-linked immuno-absorbent assay (ELISA). Normal reference ranges for MCP-1 have not been established but higher levels tend to be associated with higher body mass index.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Normal-weight | Obese
Number analyzed (Participants) | 8 | 6
pg/mL | 140.9 (37) | 160.3 (40.1)
Statistical Analysis 1: Comparison: Normal-weight vs Obese; [analysis description as in outcome 2, analysis 1]; Test type: Other — Alternative hypothesis: higher levels of MCP-1, a pro-inflammatory marker, will relate to higher levels of putative neuroinflammation in white matter tracts as measured by DBSI restricted fraction after controlling for BMI. Null hypothesis: MCP-1 levels will not be related to DBSI RF in white matter tracts after controlling for BMI; p = 0.26, Regression, Linear — a priori threshold: p < 0.05; Slope = 0.34
Statistical Analysis 2: Comparison: Normal-weight vs Obese; [analysis description as in outcome 2, analysis 1]; Test type: Other — Alternative hypothesis: higher levels of MCP-1, a pro-inflammatory marker, will relate to higher levels of putative neuroinflammation in white matter tracts as measured by DBSI hindered fraction after controlling for BMI. Null hypothesis: MCP-1 levels will not be related to DBSI HF in white matter tracts after controlling for BMI; p = 0.71, Regression, Linear — a priori threshold: p < 0.05; Slope = 0.12

11. Post Hoc Outcome: Peripheral Inflammation as Measured by Plasma Assays and Relationships With DBSI Putative Neuroinflammation Metrics in White Matter Tracts in Obese and Normal-weight Individuals
Description: Fasting plasma high-sensitive C-reactive protein (CRP), where higher levels may reflect greater low-grade inflammation. High-sensitive CRP was measured using high-sensitive CRP turbidimetry assay. Higher high-sensitive CRP levels may reflect greater risk for cardiovascular disease. Normal range for hs-CRP is usually below 1 mg/L.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Normal-weight | Obese
Number analyzed (Participants) | 8 | 6
mg/L | 1 (0.8) | 4.8 (3.1)
Statistical Analysis 1: Comparison: Normal-weight vs Obese; [analysis description as in outcome 2, analysis 1]; Test type: Other — Alternative hypothesis: higher levels of CRP, a pro-inflammatory marker, will relate to higher levels of putative neuroinflammation in white matter tracts as measured by DBSI restricted fraction after controlling for BMI. Null hypothesis: CRP levels will not be related to DBSI RF in white matter tracts after controlling for BMI; p = 0.54, Regression, Linear — a priori threshold: p < 0.05; Slope = 0.19
Statistical Analysis 2: Comparison: Normal-weight vs Obese; [analysis description as in outcome 2, analysis 1]; Test type: Other — Alternative hypothesis: higher levels of CRP, a pro-inflammatory marker, will relate to higher levels of putative neuroinflammation in white matter tracts as measured by DBSI hindered fraction after controlling for BMI. Null hypothesis: CRP levels will not be related to DBSI HF in white matter tracts after controlling for BMI; p = 0.77, Regression, Linear — a priori threshold: p < 0.05; Slope = 0.09

ADVERSE EVENTS:
Time Frame: Over one study visit, about 8 hours per participant
Arm/Group | Normal-weight | Obese
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 0/8 | 0/6

LIMITATIONS AND CAVEATS:
An early anticipated enrollment table specified a total of 8 individuals. Due to necessary change in study methods, we were able to increase the anticipated enrollment to 20 individuals. 20 individuals were enrolled but 5 met exclusion criteria during further screening (after signing informed consent) and one could not be scheduled due to scheduling conflicts (but they had signed the consent form). In total, we had complete datasets from 14 enrolled individuals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/29/NCT04116229/Prot_SAP_000.pdf